CLINICAL TRIAL: NCT02863822
Title: A Prospective, Randomized, Investigator Blinded, Controlled Trial to Evaluate the Effectiveness of Dietary Modification in Patients With Functional Dyspepsia
Brief Title: Study to Evaluate Dietary Modification in Patients With Functional Dyspepsia.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no patients enrolled
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-203
Record Dates: First submitted 2016-05-26; First posted 2016-08-11 (Estimated); Last update posted 2024-10-03 (Actual); Status verified 2018-04

CONDITIONS: Dyspepsia; Dietary Modification
Keywords: Functional Dyspepsia; Low FODMAP; Dietary Modification
MeSH Terms: conditions — Dyspepsia | interventions — FODMAP Diet

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low FODMAP (Experimental): Subjects will be given dietary education in the low FODMAP diet, which they will continue for 4 weeks. Subjects will then followup with the dietician and subjects with a symptomatic response will be given instructions for reintroduction.
  Interventions: Behavioral: Low FODMAP Diet
- Choose My Plate (Active Comparator): Subjects will receive dietary counseling in the choose my plate diet as defined by choosemyplate.gov. Subjects will also receive 2 dietician visits, 4 weeks apart.
  Interventions: Behavioral: Choose My Plate Diet

INTERVENTIONS:
Behavioral: Low FODMAP Diet — Subjects in the experimental arm, will be educated in the low fermentable oligo-di-monosaccharides and polyols (FODMAP) diet.
  Arms: Low FODMAP
Behavioral: Choose My Plate Diet — Subjects in the active comparator arm will be educated in the ChooseMyPlate.gov Diet.
  Arms: Choose My Plate

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the low fermentable oligo-di-monosaccharides and polyols (FODMAP) diet in functional dyspepsia (FD). The investigators will compare education in the low FODMAP diet to a standard healthy diet for improving symptoms in FD.

DETAILED DESCRIPTION:
Functional Dyspepsia (FD) is defined by the Rome III criteria as bothersome postprandial fullness, early satiation, epigastric pain, or epigastric burning in the absence of structural or systemic disease that can explain the symptoms. These symptoms have been present for at least 3 months with symptom onset 6 months prior to the diagnosis.

The low fermentable oligo-di-monosaccharides and polyols (FODMAP) diet has been studied in irritable bowel syndrome (IBS) patients and has been shown to have modest benefit in a limited number of small studies. The diet is generally started by complete elimination of fructose, lactose, fructans, galactans, and polyols. Following symptom improvement, these groups are reintroduced one at a time while the patient monitors for symptoms.

Although the low FODMAP diet has never been formally studied in patients with functional dyspepsia, we have noted the FD patients report improvement in their symptoms on the diet. This improvement could be explained by reduction in duodenal and gastric distention with the low FODMAP diet or a change in the duodenal flora.

To date, there have been no randomized trials evaluating dietary modification in FD. The purpose of this study is to evaluate the efficacy of the low FODMAP diet in functional dyspepsia. The investigator's hypothesis is that the addition of the FODMAP diet to standard medical treatment will result in improved symptom control in patients with functional dyspepsia.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years and older
* Diagnosis of FD with either PDS or EPS as measured by Rome III Criteria
* Patients describing inadequate relief of dyspepsia symptoms
* Endoscopy performed in the last 3 years and negative for an organic cause for dyspeptic symptoms
* H pylori negative by non-invasive testing or biopsy. Patients with a history of successfully eradicated H pylori will be included if follow-up testing by stool antigen, urea breath testing, or biopsy is negative
* Celiac disease excluded by serologies or biopsy

Exclusion Criteria:

* Patients with IBS predominant symptoms that are not well controlled
* Patients with a diagnosis of GERD who have uncontrolled heartburn
* History of esophagitis, ulcer disease, or other organic upper GI disease, including a diagnosis of celiac disease, gastroparesis, or vascular disorders of the upper GI tract
* History of surgery involving the esophagus, stomach, or duodenum
* Known lactose intolerance, unless symptoms persist on a lactose free diet
* Known fructose intolerance unless symptoms persist on a fructose free diet
* Patients undergoing active titration of any medications
* Pregnant or breastfeeding women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Self report of adequate relief | Week 7 (after 4 weeks of diet modification)
  Self report of adequate relief of dyspepsia symptoms for the previous 7 days. This information will be collected at week 7. This measure is considered clinically relevant and has been tested for responsiveness in FD

SECONDARY OUTCOMES:
Improvement in the NDI short form | Week 7 (after 4 weeks of diet modification)
  The NDI short form is a validated questionnaire used to determine the severity of symptoms related to dyspepsia. It can be used to evaluate change over time.
Improvement in the Global Overall Symptom Scale | Week 7 (after 4 weeks of diet modification)
Continued Improvement in the Global Overall Symptom Scale | Week 10 (after low FODMAP reintroduction)
Continued Improvement in the NDI short form | Week 10 (after low FODMAP reintroduction)
  The NDI short form is a validated questionnaire used to determine the severity of symptoms related to dyspepsia. It can be used to evaluate change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Hina Omar, MD, Principal Investigator — Advocate Lutheran General Hospital; Marc Fine, MD, Principal Investigator — Advocate Lutheran General Hospital
Locations (1):
- Advocate Lutheran General Hospital, Park Ridge, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
No plan to make individual participant data available. Poster presentation, Manuscript publication, oral presentations are planned.

REFERENCES:
- [Background] Staudacher HM, Lomer MC, Anderson JL, Barrett JS, Muir JG, Irving PM, Whelan K. Fermentable carbohydrate restriction reduces luminal bifidobacteria and gastrointestinal symptoms in patients with irritable bowel syndrome. J Nutr. 2012 Aug;142(8):1510-8. doi: 10.3945/jn.112.159285. Epub 2012 Jun 27. PMID 22739368
- [Background] Ong DK, Mitchell SB, Barrett JS, Shepherd SJ, Irving PM, Biesiekierski JR, Smith S, Gibson PR, Muir JG. Manipulation of dietary short chain carbohydrates alters the pattern of gas production and genesis of symptoms in irritable bowel syndrome. J Gastroenterol Hepatol. 2010 Aug;25(8):1366-73. doi: 10.1111/j.1440-1746.2010.06370.x. PMID 20659225
- [Background] Kerckhoffs AP, Samsom M, van der Rest ME, de Vogel J, Knol J, Ben-Amor K, Akkermans LM. Lower Bifidobacteria counts in both duodenal mucosa-associated and fecal microbiota in irritable bowel syndrome patients. World J Gastroenterol. 2009 Jun 21;15(23):2887-92. doi: 10.3748/wjg.15.2887. PMID 19533811
- [Background] Talley NJ, Dennis EH, Schettler-Duncan VA, Lacy BE, Olden KW, Crowell MD. Overlapping upper and lower gastrointestinal symptoms in irritable bowel syndrome patients with constipation or diarrhea. Am J Gastroenterol. 2003 Nov;98(11):2454-9. doi: 10.1111/j.1572-0241.2003.07699.x. PMID 14638348
- [Background] Talley NJ, Van Zanten SV, Saez LR, Dukes G, Perschy T, Heath M, Kleoudis C, Mangel AW. A dose-ranging, placebo-controlled, randomized trial of alosetron in patients with functional dyspepsia. Aliment Pharmacol Ther. 2001 Apr;15(4):525-37. doi: 10.1046/j.1365-2036.2001.00941.x. PMID 11284782
- [Background] Talley NJ, Locke GR, Saito YA, Almazar AE, Bouras EP, Howden CW, Lacy BE, DiBaise JK, Prather CM, Abraham BP, El-Serag HB, Moayyedi P, Herrick LM, Szarka LA, Camilleri M, Hamilton FA, Schleck CD, Tilkes KE, Zinsmeister AR. Effect of Amitriptyline and Escitalopram on Functional Dyspepsia: A Multicenter, Randomized Controlled Study. Gastroenterology. 2015 Aug;149(2):340-9.e2. doi: 10.1053/j.gastro.2015.04.020. Epub 2015 Apr 25. PMID 25921377
- [Background] Talley NJ, Verlinden M, Jones M. Quality of life in functional dyspepsia: responsiveness of the Nepean Dyspepsia Index and development of a new 10-item short form. Aliment Pharmacol Ther. 2001 Feb;15(2):207-16. doi: 10.1046/j.1365-2036.2001.00900.x. PMID 11148439